CLINICAL TRIAL: NCT00239720
Title: Treatment of Psoriatic Arthritis With hOKT3γ1 (Ala-Ala)
Brief Title: PsA Treatment With hOKT3γ1 (Ala-Ala)
Acronym: PART
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study team decision-impact(s) of change in hOKT3γ1 (Ala-Ala) manufacturer during study.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT ITN011AI
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Results first posted 2012-03-21 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-03

CONDITIONS: Arthritis, Psoriatic
Keywords: Psoriatic Arthritis; Arthritis; Psoriasis; Psoriatic; PsA
MeSH Terms: conditions — Arthritis, Psoriatic; Arthritis; Psoriasis | interventions — teplizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hOKT3gamma1 (Ala-Ala) (Experimental): Escalating dose of hOKT3gamma1 (Ala-Ala) given intravenously over 5 days of each 28 day cycle
  Interventions: Drug: hOKT3gamma1(Ala-Ala)
- Placebo (Placebo Comparator): Intravenous dose of placebo given over 5 days of each 28 day cycle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: hOKT3gamma1(Ala-Ala) — Escalating dose given IV over 5 days (1mg, 2mg, 4mg on days 3-5) of each 28 day cycle
  Other Names: anti-CD3 monoclonal antibody
  Arms: hOKT3gamma1 (Ala-Ala)
Drug: Placebo — Intravenous dose of placebo given over 5 days of each 28 day cycle
  Other Names: Placebo comparator
  Arms: Placebo

SUMMARY:
hOKT3gamma1 (Ala-Ala) is a man-made antibody that is commonly used to prevent organ rejection. The purpose of this study is to determine whether hOKT3gamma1 (Ala-Ala) is safe and effective in psoriatic arthritis patients who are unable to control their arthritis with methotrexate or azathioprine.

DETAILED DESCRIPTION:
Psoriatic arthritis is a form of inflammatory arthritis that affects approximately 7% of people who have psoriasis. Treatment typically include drugs such as methotrexate, azathioprine, and etanercept, which suppress the immune system in a nonspecific fashion in an attempt to control the immune responses causing the disease. In some severe cases of psoriatic arthritis, these drugs cannot adequately control the disease, often requiring patients to undergo continuous treatment to prevent or combat disease activity. hOKT3gamma1 (Ala-Ala) is a genetically engineered monoclonal antibody directed against the CD3 antigen on T cells. hOKT3gamma1 (Ala-Ala) specifically targets immune cells that are actively involved in destructive immune responses, such as those that cause psoriatic arthritis. In a small pilot study of eight people with psoriatic arthritis who received a 2-week course of hOKT3gamma1 (Ala-Ala), the drug appeared safe and caused no serious side effects. This study will test the safety and efficacy of hOKT3gamma1 (Ala-Ala) in alleviating symptoms in psoriatic arthritis patients.

This study will last 2 years. Individuals with psoriatic arthritis who are receiving methotrexate or azathioprine therapy and have active disease are eligible to participate. Participants will be randomly assigned to receive hOKT3gamma1 (Ala-Ala) or placebo. Participants will receive a 5-day treatment with the drug or placebo every month for the first 4 months of the study. There will be 5 study visits over 2 years to assess the safety and effectiveness of hOKT3gamma1 (Ala-Ala) and to evaluate laboratory measures related to the underlying immune problems that cause psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of psoriatic arthritis. Participants do not need to have concurrent psoriasis to participate in the study;
* Active inflammation in 3 or more joints;
* Currently receiving ongoing therapy with methotrexate or azathioprine; and
* Willing to use acceptable forms of contraception.

Exclusion Criteria:

* Active infection with HIV, hepatitis C virus, or hepatitis B virus;
* Uncompensated heart failure or a recent myocardial infarction (heart attack) within the 6 months prior to study entry;
* Certain other serious illnesses or cancers;
* Participation in another clinical trial within the 6 weeks prior to study entry; or
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-03-16 (Actual); Primary Completion 2006-12 (Actual); Study Completion 2008-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Clark, MD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - University of Colorado, Aurora, Colorado
  - University of Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Data access is provided in TrialShare, the Immune Tolerance Network (ITN) Clinical Trials Research Portal that makes data from the consortium's clinical trials publicly available.

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Immune Tolerance Network (ITN) website — http://www.immunetolerance.org
- Available data/document: Study overview, - synopsis, -navigator, -schedule of events, -available biospecimen(s) et al.: ITN011AI/NPA01 is Study ID — https://www.itntrialshare.org/project/Studies/ITN011AIPUBLIC/Study%20Data/begin.view? — TrialShare is the ITN clinical research portal that provides public access to study data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two centers in the United States enrolled four participants between March 2006 and September 2006 who had psoriatic arthritis with three or more active joints despite ongoing therapy with methotrexate or azathioprine
Pre-assignment Details: At screening visit, participants underwent procedures to establish inclusion/exclusion criteria and then sign the informed consent form
Period: Overall Study
Arm/Group | hOKT3gamma1 (Ala-Ala) | Placebo
Started | 3 | 1
Completed | 2 (One participant discontinued due to an adverse event) | 0 (One participant lost to follow-up)
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | hOKT3gamma1 (Ala-Ala) | Placebo | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (9.6) | 54 (0) | 46.3 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Received at Least Two Cycles of Treatment and Who Showed Predefined Levels of Improvement in Primary Efficacy Parameter at Six Months
Description: Participants who improve by at least 1 unit from baseline in either the physician or participant global assessment and have at least 30% improvement from baseline in either tender or swollen joint scores[1] at 6 months from start of treatment and received at least 2 cycles of treatment
  1. The tender and swollen joint scores assess 68 and 66 joints, respectively, with each joint rated from 0 to 3. Total scores range from 0-204 for tenderness and 0-198 for swelling, with higher scores indicating more severe symptoms[2].
  2. Ref: Clegg DO et al. Arthritis Rheum. 1996; 39(12):2013-20.
Time Frame: 6 Months
Population: Intent-to-treat
Arm/Group | hOKT3gamma1 (Ala-Ala) | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to end of study (up to 24 months post baseline visit)
Description: This study graded the severity of adverse events experienced by the study participant according to criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 3.0 (June 10, 2003)
Arm/Group | hOKT3gamma1 (Ala-Ala) | Placebo
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/1
Other Adverse Events (participants affected / at risk) | 2/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | hOKT3gamma1 (Ala-Ala) (N=3) | Placebo (N=1)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | hOKT3gamma1 (Ala-Ala) (N=3) | Placebo (N=1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis viral (Infections and infestations) | 1 (1) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (6) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was put on voluntary clinical hold after a serious adverse event occurred. After a review of the data, the team decided to close the study to further enrollment. Due to limited participants, no formal statistical analyses were performed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No